CLINICAL TRIAL: NCT06071650
Title: Assessment, Monitoring and Optimisation of Prehabilitation Patients Using Wearable Fitness Trackers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 308356
Record Dates: First submitted 2023-08-31; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Cancer
Keywords: preoperative exercise; prehabilitation; activity tracker; kinesiotherapy
MeSH Terms: conditions — Neoplasms | interventions — Fluconazole

STUDY DESIGN:
Intervention Model Description: A prospective, two-arm randomised parallel group clinical trial. Prehabilitation is routinely offered as the standard of care to all patients who are scheduled for curative resectional surgeries for upper gastrointestinal (UGI) cancer at Imperial College Healthcare Trust and lung cancer at Guy's and St Thomas' NHS Foundation Trust.
  Consecutive patients referred for prehabilitation will be approached for enrolment into the study. If willing to participate, written informed consent will be gained (e-consent). Following enrolment all participants will be provided with a wearable fitness tracker and will be randomised to one of two groups (1:1 randomisation) - Group A or Group B. The only difference between the two groups is the prescription of exercise, all other activities and data collected are the same.
  Randomisation following recruitment and using a computer programme.
Masking Description: Because of the nature of the study and the interventions offered, it will not be possible to blind participants or research assistants to allocation groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Exercise to Rating of Perceived Exertion (RPE) - "Control Group" (No Intervention): Participants prescribed moderate intensity aerobic exercise using their rating of perceived exertion (RPE) with a goal of sustaining an intensity level of 12 to 14 for their prescribed duration.
- Group B - Exercise to a Heart Rate (HR) Zone - "Intervention Group" (Experimental): Participants prescribed moderate intensity aerobic exercise using personalised heartrate zones with a goal of sustaining an intensity level by maintaining their heartrate above 50 percent of their heartrate reserve level for their prescribed duration.
  Interventions: Behavioral: Exercise to a Heart Rate (HR) Zone

INTERVENTIONS:
Behavioral: Exercise to a Heart Rate (HR) Zone — Participants prescribed moderate intensity aerobic exercise using personalised heartrate zones with a goal of sustaining an intensity level by maintaining their heartrate above 50 percent of their heartrate reserve level for their prescribed duration
  Arms: Group B - Exercise to a Heart Rate (HR) Zone - "Intervention Group"

SUMMARY:
Prehabilitation is the use of exercise prior to surgery to improve peoples' fitness, which leads to improved outcomes of surgery. This service is now being run remotely, however, there is little existing evidence to support the best practice for this. Currently, baseline fitness is assessed remotely using either a sit to stand test or a step test. Once completed people are prescribed regular exercises and asked to exercise to a level of intensity using a measure called Rating of Perceived Exertion (RPE). However, these measurements may not be reliable. We are carrying out a study to assess if another waking test (modified Rockport test) and asking patients to exercise to a target heart rate are better measures of assessing baseline fitness and exercise intensity.

All participants will receive weekly telephone calls to check their progress and be provided with a wrist worn fitness tracker (Fitbit). Participants will be randomised to one of two groups. The only difference between the groups will be the way the exercise is prescribed. In one group participants will be asked to complete the exercises to an exercise level they find "somewhat hard". The other group will be asked to complete the exercises to maintain a set heart rate.

All participants will be asked to complete an activity log (submitted weekly) as an online form. A small group of people (maximum 10) will be asked if they would like to complete an in-person baseline fitness assessment also, this is optional.

This study runs for up to eight weeks with participation ending after eight weeks or at the time of surgery, whichever is sooner. In the final week of participation, participants will be asked to complete an online questionnaire about their experience of using a wearable fitness tracker during the prehabilitation programme.

DETAILED DESCRIPTION:
Optimising patients pre-operatively or "Prehabilitation" is a relatively new and evolving concept in patient care. Prehabilitation utilises prescribed exercise in the time prior to surgery with the aim of improving a patient's functional capacity enabling them to better withstand the stress of surgery. 1-3 This is required due to the physiological insult cause by surgery, particularly in those with cancer, which in turn results in a decline in patients' function.

Post-operative restorative rehabilitation programmes such as Enhanced Recovery After Surgery (ERAS) are commonplace and used with the aim of returning the patients' function towards their preoperative baseline. ERAS has been shown to improve postoperative outcomes, including length of stay, re-admission, and complication rates.4 Prehabilitation has been shown to both improve cardiovascular fitness prior to surgery5,6 and like ERAS reduce post-operative complications.7,8 However, despite this and unlike ERAS, it's use is still patchy, with no national protocols in existence.

Due to evidence demonstrating its effectiveness, the benefits of commissioning prehabilitation services have been acknowledged in several surgical fields,9 with national policy documents from NHS England placing an emphasis on preventative rehabilitation, delivered before and during cancer treatment.10 As such, the policy environment could be seen as favourable. However, there is little evidence available, and significant heterogeneity in that which is available, for how best to approach a prehabilitation service to achieve the best results.

Physical activity is a core component seen across all reported prehabilitation programmes. However, heterogeneity is seen across multimodal programmes, meaning the type of exercise, duration and supervision of physical activity is inconsistently administered between studies. Additional interventions such as dietary support, psychological wellbeing and smoking cessation are also variably addressed in some studies.

Accurate, reliable, and reproducible assessment of cardiopulmonary fitness is required to effectively prescribe and monitor patients as they progress through a prehabilitation programme. Currently, cardiopulmonary fitness assessment requires patients to attend for in person assessment to undergo Maximal or Submaximal exercise testing.

WEARABLE ACTIVITY TRACKING AND EHEALTH TECHNOLOGIES IN HEALTHCARE

Wearable "fitness tracking" technologies incorporating sensors which monitor activity and physiological parameters are now pervasive and are a rapidly expanding commercial industry worldwide with a market size valuation of USD 37.10 billion in 2020, and a projected compound annual growth rate of 15.9% from 2020 to 2027.11 With significant investment in this technology leading to increasing functionality, reliability and aesthetics it opens up the potential for use in a healthcare setting where to date their use has already been shown to be both feasible and insightful in the perioperative setting.12 Intuitively, these devices could provide a beneficial aid in prehabilitation programmes. However, a literature review found no studies have yet reported the use of wearable technologies on patients when used within a prehabilitation programme.

eHealth technologies are defined as the cost-effective and secure use of information and communications technologies in support of health and health-related fields13. They are already widely used by patients with 72% of internet users saying they looked online for health information of one kind or another within the past year14 and 69% of adults regularly tracking a health indicator like weight, diet, exercise routine, or symptom15. Utilising eHealth technology within prehabilitation may help to improve patient participation, particularly in home-based programmes. The assessment of exercise intensity is one possible area in which it could be used to overcome the limitations of self-assessment. Making it easier for patients to assess intensity and monitor the frequency that they are achieving their target activity may improve exercise behaviour and consequently improve the response to prehabilitation.

RATIONALE FOR CURRENT STUDY

Using fitness trackers in prehabilitation opens up the potential for remote programmes whilst maintaining objective measurement of heart rate and step count. Remote prehabilitation programmes, as opposed to in person individual or group sessions within a hospital setting are attractive to patients, health professionals and policy makers alike. For patients, the distance from home and the physical and financial demands of travel can negatively impact accessibility of programmes and the time available to complete exercises. Particularly pertinent for those travelling long distances to tertiary centres for cancer treatment and more recently with the risks of COVID-19 to those clinically vulnerable. Therefore, reducing unnecessary hospital visits is desirable. Remote assessment makes scheduling easier for clinicians and the use of wearable fitness trackers provides a more detailed understanding of individual parameters over longer periods, rather than a snapshot. For policy makers, remote assessment means reduced clinic and or gym space required, therefore reducing costs and reduced footfall (a key target resulting from the covid-19 pandemic) within the hospital to facilitate other scheduling commitments. Whilst many perceived benefits exist, it is also necessary to acknowledge that the use of fitness trackers and remote assessment may not benefit all, an area which will be addressed in this work. Whilst many remote programmes do now exist, the use of fitness trackers to support these programmes has not been assessed.

Exercise intensity Many reported programmes use a measure called Rating of Perceived Exertion (RPE) to measure exercise intensity. RPE is a widely used and validated scale that has been shown to accurately correspond to intensity measured by maximum heart rate (HRmax) in many different populations.16-18 However, as a self-reported measure, it is inherently prone to measurement bias; a preliminary study found that over 60% of RPE measurements made by patients during prehabilitation were overestimates of the actual achieved intensity measured by achieved heart rate. It is therefore proposed that using fitness trackers individuals could exercise to prescribed heart rate zones to improve achievement of their exercise targets. A heart rate zone is a range of heart rates which corresponds to a desired training effect for an individual. They can be calculated as a percentage of the heart rate reserve (HRR) which is the maximum heartrate (HRmax) an individual can achieve minus their resting heartrate (RHR).

Existing prehabilitation programs prescribe the intensity of aerobic exercises to patients by asking them to exercise to a rating of perceived exertion (RPE). As a self-reported measure, there is an inherent propensity towards measurement bias, with studies reporting over 60% of RPE measurements made by patients during prehabilitation as overestimates of the actual intensity achieved when measured by their heart rate. Therefore, I hypothesise that prescribing to a heart rate zone and providing a heart rate tracker to monitor this will increase the levels of moderate intensity exercise achieved.

Self-reporting and Adherence

Direct links have been reported between the amount of physical activity completed each week and post operative outcomes (lower risk of post-operative pneumonia with increasing volumes of activity completed in the pre-operative period). 19 However, current programmes are reliant on self-reported adherence, making assessment of the true benefits challenging. A previous study of the PREPARE programme found an average adherence of 64% to the prescribed exercise.20 Adherence to home-based exercises is often lower than supervised programmes 21 and exercise participation during chemotherapy is particularly challenging.22 It is therefore important to explore ways to remotely support and encourage patients to follow their exercise programmes during prehabilitation. Fitness trackers provide a potential objective measurement of adherence to prescribed targets.

It is beneficial to provide home (vs. hospital) based exercise programmes. However, their effectiveness dependent on patients' adherence to the prescribed physical exercises (currently self-reported via an activity log), where activity is frequently over-reported. Heart rate trackers provide data on activity level and therefore can be used remotely to determine compliance.

Patient satisfaction of using fitness trackers

Whilst the theory of using fitness trackers in remote prehabilitation is attractive, it is only beneficial if the target population are engaged, willing and able to use the devices for the desired purposes. It is important to acknowledge that the demographics of those undertaking prehabilitation for OG, HPB and LC resections may not be representative of the average and could find the use of these technologies challenging.

There is no current evidence to demonstrate that patients find the use of wearable fitness trackers in prehabilitation acceptable. The benefits of using wearable fitness trackers in prehabilitation will be reduced if compliance with the device is low (i.e., they do not wear them). Therefore, there is a need to assess the acceptability, usability, and user experience of using heart rate trackers in a prehabilitation setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years.
* New diagnosis of non-metastatic oesophago-gastric (OG), hepatobiliary (HPB) or Lung Cancer (LC) being offered surgical resection with curative intent at Imperial College NHS Healthcare Trust (OG/HPB) or Guy's and St Thomas' Hospital (LC).
* Proficient in English
* Enrolled in a prehabilitation programme.
* Capable of providing informed consent and willing to comply with all parts of the protocol.

Exclusion Criteria:

* Unable to provide informed consent.
* Non-resectable disease.
* Declined surgery.
* No access to smart phone/tablet or internet
* Involved in other current research or have recently been involved in any research prior to recruitment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Total number of minutes of moderate intensity exercise | Data collected from each participant for up to 8 weeks or until they have undergone their cancer resection. The end of the study will be on completion of data collection from the 82nd participant.
  The primary outcome will compare between intervention and control groups the total number of minutes of moderate intensity exercise, i.e., exercise within target range as measure on the Fitbit over the 8 weeks of follow-up

SECONDARY OUTCOMES:
Volume of physical activity (mean MET min/week) achieved. | Data collected from each participant for up to 8 weeks or until they have undergone their cancer resection. The end of the study will be on completion of data collection from the 82nd participant.
  A comparison of the volume of physical activity (mean MET min/week) achieved between the intervention and control groups over the 8 weeks of follow-up.
Weekly adherence (mean percentage of actual/prescribed MET minutes/week) | Data collected from each participant for up to 8 weeks or until they have undergone their cancer resection. The end of the study will be on completion of data collection from the 82nd participant.
  A comparison of weekly adherence (mean percentage of actual/prescribed MET minutes/week) between the intervention and control groups over the 8 weeks of follow-up.
Duration of exercise self-reported vs recorded HR data (minutes) | Data collected from each participant for up to 8 weeks or until they have undergone their cancer resection. The end of the study will be on completion of data collection from the 82nd participant.
  Comparison between participants self-reported duration of exercises (minutes) and their recorded duration of achieving >40% of their heart rate reserve (minutes).
Intensity of exercise self-reported vs recorded HR data (RPE vs % of target HR zone) | Data collected from each participant for up to 8 weeks or until they have undergone their cancer resection. The end of the study will be on completion of data collection from the 82nd participant.
  Comparison between participants self-reported intensity of exercises and their recorded heart rate intensity data (RPE vs % of target HR zone achieved) .
Patient feedback of using heart rate trackers in a prehabilitation setting - Technology acceptance Model (TAM) | Questionnaire collected from each participant at the end of their heart rate data collection (after 8 weeks or until they have undergone their cancer resection)
  Descriptive analysis assessing the acceptability of the intervention to the participants using a validated questionnaire at the end of the intervention period.
  TAM - 12 questions (6 on perceived usefulness. 6 on perceived Ease-of-use) each graded on a 7 point Likert scale
Patient feedback of using heart rate trackers in a prehabilitation setting - UMUX-lite | Questionnaire collected from each participant at the end of their heart rate data collection (after 8 weeks or until they have undergone their cancer resection)
  Descriptive analysis of a validated questionnaire assessing usability of the intervention to the participants taken at the end of the intervention.
  UMUX-lite - 2 questions graded on a 7 point Likert scale
Patient feedback of using heart rate trackers in a prehabilitation setting - UEQ | Questionnaire collected from each participant at the end of their heart rate data collection (after 8 weeks or until they have undergone their cancer resection)
  Descriptive analysis of the participants user experiences of the intervention using a validated questionnaire at the end of the intervention.
  UEQ - 26 pairs of contrasting attributes that may apply to the product each to be graded on a 7 point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Moorthy, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No